CLINICAL TRIAL: NCT07144943
Title: Study on the Observation of the Evolution of Sexual Symptoms in Sexual Offenders With Paraphilia (With or Without Antiandrogen or SSRI Treatments)
Brief Title: "Evolution of Sexual Symptoms in Paraphilic Sexual Offenders With/Without Antiandrogen or SSRI Treatment"
Acronym: ESPARA
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier St Anne (Other)
Responsible Party: Sponsor
Other Study IDs: D24-P008; 2024-A01543-44 (Other: ANSM)
Record Dates: First submitted 2025-08-04; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Sexual Disorder, Physiological
Keywords: sexual offenders; paraphilia; ESPARA
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Paraphilic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- patients on antiandrogens: standard care
  Interventions: Radiation: For subjects on SSRIs: bone densitometry
- patients on SSRI: selective serotonin reuptake inhibitors
  Interventions: Radiation: For subjects on SSRIs: bone densitometry
- patient without pharmacological treatment

INTERVENTIONS:
Radiation: For subjects on SSRIs: bone densitometry — For subjects on SSRIs:
  Bone densitometry is one of the additional examinations considered. This assessment is part of the routine monitoring for subjects on androgens.
  Other Names: patients on SSRIs
  Groups: patients on SSRI; patients on antiandrogens

SUMMARY:
The ESPARA study is a multicenter observational research project aiming to monitor, over a three-year period, the evolution of sexual symptoms in male sexual offenders with paraphilia, divided into three groups: receiving antiandrogen treatment, receiving selective serotonin reuptake inhibitors (SSRIs), or no pharmacological treatment. The primary objective is to assess changes in sexual desire intensity and deviant sexual behaviors, while secondary objectives include relapse rates, the role of psychiatric comorbidities, treatment tolerability, and various clinical, cognitive, and life-history factors.

DETAILED DESCRIPTION:
This is a prospective longitudinal cohort study including 200 male participants aged 18-65 years, diagnosed with a paraphilic disorder according to DSM-5, and convicted of sexual offenses (e.g., exhibitionism, rape, sexual assault, incest, possession of child sexual abuse material). Participants are recruited in their usual care setting, after providing informed consent, and assigned to one of three cohorts based on current treatment: antiandrogens, SSRIs, or no pharmacological treatment.

Over a 3-year follow-up period, participants undergo standardized assessments every 3 months, including:

Measurement of sexual desire intensity and deviant sexual symptoms (validated self-report scales).

Recording of any relapses (self-reported, third-party notifications). Evaluation of psychiatric comorbidities (DSM-5), personality disorders (PDQ-4+), impulsivity (BIS-11), and treatment adherence (BARS).

Biological analyses (testosterone levels and others) and regular clinical examinations.

Cognitive and psychological assessments (empathy, denial, cognitive distortions, hypersexuality, alcohol/drug use).

Documentation of traumatic life events (THQ). Optional genetic study through saliva and blood sampling. The study does not initiate or modify treatment; all medical decisions remain under the responsibility of the treating physician. Any adverse effects are systematically documented. Data will be analyzed within each group and, when appropriate, compared between groups after statistical adjustment.

The project is funded by a national PHRC grant and has received ethics committee approval. Additional risks for participants are considered minimal, as all assessments and examinations align with standard care practices.

ELIGIBILITY:
Inclusion Criteria:

* Men suffering from paraphilias (DSM-5 criteria),
* Aged 18 to 65 years,
* Sexual offenders (offense or sexual assault including exhibitionism, rape, sexual touching, incest, possession of pedopornographic video material) (severity level 1 to 6 according to WFSBP recommendations),
* Subject who has given consent,
* Patients covered by social security,
* Satisfactory command of written and spoken French."

Exclusion Criteria:

* Subject in prison (regardless of the reason),
* Subject under guardianship (patients under legal supervision may, however, be included),
* Subjects who have committed a sexual offense and do not meet the DSM-5 criteria for paraphilia."

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: * Men suffering from paraphilic disorders (DSM-5 criteria),
  * Aged between 18 and 65 years,
  * Sexual offenders (offense or sexual assault including exhibitionism, rape, sexual touching, incest, possession of child pornographic video material) (severity level 1 to 6 according to WFSBP guidelines)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Change in sexual desire and paraphilic behavior scores using the Intensity of Sexual Desire and Sexual Symptoms Scale (ISDSS, self-report) | Baseline
  The ISDSS assesses three domains of sexual functioning during the past month:
  Sexual interest and desire (score 0-8; higher = stronger desire)
  Sexual thoughts and fantasies (score 0-8; higher = more frequent/intense fantasies)
  Frequency of paraphilic sexual activities per week (e.g., masturbation, sexual activity leading to orgasm; reported as count).
  The mean score of the three domains (range 0-8) will be calculated. Higher scores indicate worse outcome (greater intensity/frequency of paraphilic sexual behavior).

SECONDARY OUTCOMES:
Sexual relapse occurrence | 3 months
  Number of participants with sexual relapse (recurrence of deviant sexual behavior) during the 36-month follow-up, recorded at each 3-month visit via participant report, third-party notifications, or official records.
Presence of psychiatric disorders according to DSM-5 criteria | Baseline and 36 months.
  Categorical diagnosis (present/absent) of psychiatric comorbidities assessed at baseline and 36 months using the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria.
Change in treatment adherence - Brief Adherence Rating Scale | 3 months
  Outcome: Change from baseline in treatment adherence score at 36 months. Measurement: Measured every 3 months using the Brief Adherence Rating Scale (BARS, range 0-6; higher scores indicate better adherence).
Treatment-related adverse events | At baseline
  Number of participants with treatment-related adverse events during the 36-month follow-up, documented by type, frequency, onset time, and severity, as reported by the treating physician or participant.
Presence of clinically observable gynecomastia | 3 months.
  Binary assessment (present/absent) of gynecomastia at baseline and every 3 months.
Traumatic life events (THQ - Trauma History Questionnaire) | At baseline
  Outcome: Total score on the Trauma History Questionnaire (THQ). Measurement: THQ is a self-report questionnaire assessing the presence and frequency of traumatic events over the lifetime.
  Scale: The French version used in the study includes a series of items scored from 0 (no occurrence) to a maximum determined by the number of events endorsed (higher scores indicate a greater number of traumatic events).
  Scoring interpretation: Higher scores reflect a worse outcome, meaning greater exposure to traumatic life events.
Change in clinical management - Comorbidity | 3 months
  Number of participants whose comorbidity profile changes during the 36-month follow-up.
  Measurement: Recorded at each 3-month visit, based on DSM-5 diagnosis status (present/absent for each condition
Change in clinical management - Treatment tolerance | 3 months
  Number of participants with changes in clinical management due to treatment-related adverse events.
  Measurement: Recorded at each 3-month visit; events classified by type, severity, and relationship to treatment (CTCAE v4.0).
Change in clinical management - Sexual symptoms evolution | 3 months
  Outcome: Change from baseline in sexual symptom scores leading to a modification of clinical management.
  Measurement: Difference in scores from validated sexual symptoms scales (libido, fantasies, sexual activity), measured every 3 months over 36 months.
Change in treatment adherence - Serum testosterone level | At 36 months
  Outcome: Change from baseline in serum testosterone concentration at 36 months in participants receiving SSRIs or antiandrogens.
  Measurement: Measured in ng/dL at baseline and when non-adherence is suspected; lower levels are expected in adherent participants on antiandrogen treatment.
Personality traits measured with the Personality Diagnostic Questionnaire-4+ (PDQ-4+) | Baseline and 36 months.
  The PDQ-4+ assesses personality disorder traits. Score range 0-100; higher scores indicate more personality disorder traits (worse outcome).
Impulsivity measured with the Barratt Impulsiveness Scale, Version 11 (BIS-11) | Baseline and 36 months.
  The BIS-11 is a self-report questionnaire of impulsivity. Score range 30-120; higher scores indicate greater impulsivity (worse outcome).
Change in systolic and diastolic blood pressure (mmHg) | 3 months.
  Mean systolic and diastolic blood pressure values measured at baseline and every 3 months.
Change in body weight (kg) | 3 months.
  Mean weight measured at baseline and every 3 months.
Aggression measured with the Molest Scale | 3 months.
  Description: Molest Scale score, range [min-max to be specified], higher scores indicate greater aggression (worse outcome).
Sexual violence risk measured with the Rape Scale | 3 months.
  Rape Scale score, range [min-max], higher scores indicate higher risk of sexual violence (worse outcome).
Empathy score [specify full name of empathy scale] | 3 months.
  Range [min-max], higher scores indicate greater empathy (better outcome).
Denial score [specify full name of denial scale] | 3 months.
  Range [min-max], higher scores indicate greater denial (worse outcome).
Alcohol use measured with the Alcohol Use Disorders Identification Test (AUDIT) | 3 months.
  AUDIT total score (0-40). Higher scores indicate more hazardous or harmful drinking (worse outcome).
Illicit drug use (type, quantity, duration) | 3 months.
  Self-reported consumption of illicit drugs (type, grams/day, duration). Reported at baseline and every 3 months.
Hypersexuality screening with PATHOS and PEACCE | 3 months.
  PATHOS score range 0-5, PEACCE [specify range]. Higher scores indicate higher risk of hypersexuality (worse outcome).
Compulsive sexual behavior measured with the Compulsive Sexual Behavior Inventory (CSBI) | 3 months.
  CSBI score range [min-max], higher scores indicate greater compulsive sexual behavior (worse outcome).
Sexual violence risk measured with the STATIC-99 | 3 months.
  STATIC-99 score range 0-12; higher scores indicate greater risk of sexual violence recidivism (worse outcome).
Sexual risk factors measured with the STABLE-2007 | 3 months.
  STABLE-2007 score range 0-26; higher scores indicate greater dynamic risk factors for sexual recidivism (worse outcome).
Cognitive function measured with the Montreal Cognitive Assessment (MoCA) | Baseline
  MoCA score range 0-30; higher scores indicate better cognitive function.
Cognitive flexibility measured with the Stroop Test | Baseline
  Stroop performance (reaction time in seconds and number of errors). Longer reaction times and more errors indicate worse cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Florence THIBAUT, Professor, Principal Investigator

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (3):
  • Study Protocol (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT07144943/Prot_000.pdf
  • Informed Consent Form: Consentement éclairé pour patient majeur (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT07144943/ICF_001.pdf
  • Informed Consent Form: Consentement éclairé pour patient sous curatelle (2025-02-07): https://cdn.clinicaltrials.gov/large-docs/43/NCT07144943/ICF_002.pdf